CLINICAL TRIAL: NCT05420155
Title: Outcome After Surgical Treatment of Liver Hydatid Cyst
Brief Title: Surgical Treatment of Liver Hydatid Cyst (SURGHIDA)
Acronym: SURGHIDA
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Collaborators: Complejo Hospitalario Universitario de Badajoz (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Profesor, Universidad de Extremadura
Other Study IDs: UE-CHUB-001-2022
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Echinococcosis, Hepatic
MeSH Terms: conditions — Echinococcosis, Hepatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical group: Patients operated on liver hydatidic cyst
  Interventions: Procedure: Surgical resection

INTERVENTIONS:
Procedure: Surgical resection — Surgical treatment of hepatic hydatidic cyst

SUMMARY:
The aim was to analyses the incidence and the independent factors associated with Textbook Outcome following surgical treatment of liver hydatid cysts (LHC).

DETAILED DESCRIPTION:
Textbook outcome (TO) is a composite measure to determine the ideal postoperative period and to assess the quality of surgical care. The aim was to analyses the incidence and the independent factors associated with TO following surgical treatment of liver hydatid cysts (LHC).

The investigators conducted a retrospective cohort study of patients operated on for hepatic hydatidosis between January 2006 to December 2021. TO occurred when all the following criteria were fulfilled: no mortality within 90 days, no major complications within 90 days, no reintervention within 90 days and no prolonged hospital stay. Univariable and multivariable analyses were performed to identify factors associated with TO.

ELIGIBILITY:
Inclusion Criteria:

* Patients with liver hydatid cyst treated by total or partial pericystectomy

Exclusion Criteria:

* emergency surgery and simple drainage of cyst

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver hydatid cyst (LHC) diagnosed by preoperative computed tomography (CT) or magnetic resonance imaging (MRI) and pathological diagnosis after surgery, treated by total or partial pericystectomy
Sampling Method: Non-Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 90 days
  no mortality within 90 days
Morbidity | 90 days
  no major complications within 90 days
Re-admission | 90 days
  no re-admissions within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Gerardo Blanco-Fernández, MD, PhD, Study Director — University of Extremadura

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manterola C, Otzen T, Urrutia S; MINCIR Group (Methodology and Research in Surgery). Risk factors of postoperative morbidity in patients with uncomplicated liver hydatid cyst. Int J Surg. 2014;12(7):695-9. doi: 10.1016/j.ijsu.2014.05.063. Epub 2014 May 21. PMID 24859488
- [Background] van Roessel S, Mackay TM, van Dieren S, van der Schelling GP, Nieuwenhuijs VB, Bosscha K, van der Harst E, van Dam RM, Liem MSL, Festen S, Stommel MWJ, Roos D, Wit F, Molenaar IQ, de Meijer VE, Kazemier G, de Hingh IHJT, van Santvoort HC, Bonsing BA, Busch OR, Groot Koerkamp B, Besselink MG; Dutch Pancreatic Cancer Group. Textbook Outcome: Nationwide Analysis of a Novel Quality Measure in Pancreatic Surgery. Ann Surg. 2020 Jan;271(1):155-162. doi: 10.1097/SLA.0000000000003451. PMID 31274651
- [Background] de la Plaza Llamas R, Ramia Angel JM, Bellon JM, Arteaga Peralta V, Garcia Amador C, Lopez Marcano AJ, Medina Velasco AA, Gonzalez Sierra B, Manuel Vazquez A. Clinical Validation of the Comprehensive Complication Index as a Measure of Postoperative Morbidity at a Surgical Department: A Prospective Study. Ann Surg. 2018 Nov;268(5):838-844. doi: 10.1097/SLA.0000000000002839. PMID 30303875
- [Background] Mehta R, Tsilimigras DI, Pawlik TM. Assessment of Magnet status and Textbook Outcomes among medicare beneficiaries undergoing hepato-pancreatic surgery for cancer. J Surg Oncol. 2021 Sep;124(3):334-342. doi: 10.1002/jso.26521. Epub 2021 May 7. PMID 33961716
- [Background] Jaen-Torrejimeno I, Lopez-Guerra D, Prada-Villaverde A, Blanco-Fernandez G. Pattern of Relapse in Hepatic Hydatidosis: Analysis of 238 Cases in a Single Hospital. J Gastrointest Surg. 2020 Feb;24(2):361-367. doi: 10.1007/s11605-019-04163-7. Epub 2019 Feb 26. PMID 30809783